CLINICAL TRIAL: NCT03927651
Title: Intraoperative Use of Intravenous Indocyanine Green (ICG) to Assess Ovarian Perfusion Using Infrared Imaging: A Feasibility Pilot Study
Brief Title: ICG to Assess Ovarian Perfusion
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Magdy Milad, MD, Chief of Minimally Invasive Gynecologic Surgery in the Department of Obstetrics and Gynecology Albert B. Gerbie, MD, Professor of Obstetrics and Gynecology Professor of Obstetrics and Gynecology (Minimally Invasive Gynecologic Surgery), Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: STU00208846
Record Dates: First submitted 2019-04-09; First posted 2019-04-25 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Fibroid Uterus; Endometriosis; Uterus Myoma; Uterine Fibroid; Uterine Adenomyosis; Endometrial Cyst; Uterine Cyst
MeSH Terms: conditions — Leiomyoma; Endometriosis; Myofibroma; Adenomyosis | interventions — Indocyanine Green

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Administration of ICG (Experimental): ICG will be injected intravenously to assess ovarian perfusion in the presence or absence (control) of pathology. Near infrared fluorescence imaging will be used to illuminate the ICG. The extent of perfusion will be determined using digital imaging software. ICG will be stored at the NM Investigational Pharmacy and administered intravenously by the anesthesiologist at the direction of the surgeon during surgical procedure.
  Interventions: Drug: ICG

INTERVENTIONS:
Drug: ICG — Indocyanine green (ICG) is a Food and Drug (FDA)-approved tricarbocyanine dye that is fluorescent under near-infrared (NIR) light. ICG solutions for injection often contain sodium iodide. ICG is water soluble and when introduced intravenously, it is bound by plasma proteins, namely albumin. The intravascular half-life of ICG is 3-4 minutes with rapid hepatic clearance.
  Other Names: Indocyanine green (ICG)

SUMMARY:
To assess the feasibility of using intravenous ICG to characterize the vascular perfusion of ovaries during gynecologic surgery

DETAILED DESCRIPTION:
The purpose of this study is to determine the feasibility of intravenous ICG administration to facilitate assessments of ovarian vascular perfusion. Historically, assessment of ovarian perfusion has been performed visually or via ultrasound with Doppler evaluation. In patients with ovarian endometriomas, evidence of ovarian interstitial microvascular injury has been demonstrated similarly by the presence of low flow and high RI. The use of ICG to evaluate ovarian perfusion specifically has not been reported. The use of ICG for intraoperative perfusion assessment of the ovary could provide more information about the health of the ovary and inform the surgical approach to ovarian pathology.

ICG will be injected intravenously to assess ovarian perfusion in the presence or absence (control) of pathology. Near infrared fluorescence imaging will be used to illuminate the ICG. The extent of perfusion will be determined using digital imaging software.

ELIGIBILITY:
Inclusion Criteria:

* Patients attending a preoperative visit at the Center for Comprehensive Gynecology who will undergo surgery.

Exclusion Criteria:

* Not able to comprehend and sign a written consent
* Patients with a history of allergy to iodides
* Patients history of renal failure or uremia, and those on dialysis

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2022-11-15 (Actual); Study Completion 2022-11-15 (Actual)

PRIMARY OUTCOMES:
Assessment of ovarian perfusion after ICG administration via fluorescent imaging | 2 years
  The investigators will be assessing the feasibility of using intravenous ICG to characterize the vascular perfusion of ovaries by imaging. During surgery ICG will be administered intravenously via a peripheral or central line at the direction of the surgeon by the anesthesiologist. The injected amount will be a 3 mL solution of reconstituted ICG that contains a 7.5 mg dose of ICG. This will be followed by a 10 mL bolus of normal saline for injection per the manufacturer's recommendation. The total dose of dye injected should not exceed 2 mg/kg.
  Visibility of the ICG fluorescence should occur within 1-2 minutes with a duration of 20-120 minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Magdy Milad, MD,MS, Principal Investigator — Northwestern University
Locations (1):
- 259 E Erie - Northwestern, Chicago, Illinois, United States

DOCUMENTS (2):
  • Study Protocol (2020-06-08): https://cdn.clinicaltrials.gov/large-docs/51/NCT03927651/Prot_000.pdf
  • Informed Consent Form (2020-06-08): https://cdn.clinicaltrials.gov/large-docs/51/NCT03927651/ICF_001.pdf